CLINICAL TRIAL: NCT00411697
Title: Assess Long-term Persistence of Hepatitis B Antibodies & Immune Response to a Hepatitis B Vaccine (Engerix-B Kinder) Challenge in Children Aged 4-5 Years (Previously Primed & Boosted in the 1st 2 Years of Life With DTPa-HBV-IPV/Hib Vaccine)
Brief Title: Persistence of Hepatitis B Antibody Levels & Immune Response to a Hepatitis B Vaccine Challenge
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 106789
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

ARMS (1):
- Group A (Experimental)
  Interventions: Biological: Engerix™-B Kinder

INTERVENTIONS:
Biological: Engerix™-B Kinder — Intramuscular injection, 1 dose

SUMMARY:
The purpose of this study is to determine at 5 years of age the persistence of immunity to hepatitis B that was conferred by infant vaccination with Infanrix hexa™.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol
* A male or female of 4 to 5 years of age at the time of enrolment.
* With documented evidence of previous vaccination with four consecutive doses of Infanrix hexa™ in Germany.
* Written informed consent obtained from the parents or guardians of the subject at the time of enrolment.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product .
* Evidence of previous hepatitis B booster vaccination since administration of the fourth dose of Infanrix hexa™ booster in the second year of life.
* History of or intercurrent hepatitis B disease.
* Hepatitis B vaccination at birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before booster vaccination and ending 30 days after.
* Administration of immunoglobulins and/or any blood products within the three months preceding booster vaccination or planned administration during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the HBV vaccine challenge.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Anti-hepatitis B surface antigen (HBs) antibody concentrations | One month after the challenge dose of HBV vaccine

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | Before and after challenge dose of HBV vaccine
Occurrence of serious adverse events | During the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- Germany (28):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bietigheim-Bissingen, Baden-Wurttemberg
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Ehingen, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Herbolzheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Kirchzarten, Baden-Wurttemberg
  - GSK Investigational Site, Oberstenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Pforzheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tettnang, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Tegernsee, Bavaria
  - GSK Investigational Site, Dudenhofen, Rhineland-Palatinate
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Gau-Odernheim, Rhineland-Palatinate
  - GSK Investigational Site, Gerolstein, Rhineland-Palatinate
  - GSK Investigational Site, Schoeneberg - Kuebelberg, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Steiner M, Ramakrishnan G, Gartner B, Van Der Meeren O, Jacquet JM, Schuster V. Lasting immune memory against hepatitis B in children after primary immunization with 4 doses of DTPa-HBV-IPV/Hib in the first and 2nd year of life. BMC Infect Dis. 2010 Jan 15;10:9. doi: 10.1186/1471-2334-10-9. PMID 20078876
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 106789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register